CLINICAL TRIAL: NCT01697384
Title: Phase III, Open-Label Study to Evaluate Efficacy and Safety of Histrelin Subdermal Implant in Patients With Advanced Prostate Cancer
Brief Title: Study to Evaluate Efficacy and Safety of Histrelin Subdermal Implant in Men With Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301
Record Dates: First submitted 2011-07-13; First posted 2012-10-02 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate
Keywords: prostate cancer, PSA
MeSH Terms: conditions — Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic | interventions — histrelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one histrelin acetate 50 mg implant (Experimental): The test product was a histrelin acetate 50 mg hydrogel implant surgically placed subdermally into the inner aspect of the upper arm.
  Interventions: Drug: histrelin acetate

INTERVENTIONS:
Drug: histrelin acetate — 52 week implant
  Other Names: Vantas

SUMMARY:
Objective was to evaluate the efficacy and safety of the histrelin acetate subdermal implant (originally versus Lupron Depot-3 Month) in male patients with advanced prostate cancer during 52 weeks of treatment with the implant. After consultation w/ FDA, design was modified to eliminate the Lupron arm and continued the study as an open-label non-randomized study.

Primary endpoint was testosterone suppression, as assessed by the percent of patients whose testosterone indicated chemical castration levels (<=50 ng/dL) through 52 weeks of treatment with an implant.

DETAILED DESCRIPTION:
Other outcome measures included serum levels of LH, PSA, as well as non-clinical assessments, eg, WHO Performance Status, pain level assessment, and quality of life questionnaires. Safety was evaluated via adverse events, vital signs, clinical laboratory outcomes, physical examinations, and ECGs. Local tolerability outcomes were also evaluated.

An extension period for the study included annual replacement of the implant until the implant was approved by the FDA (October 12, 2004). Efficacy and safety were followed during the extension period.

ELIGIBILITY:
Key Inclusion Criteria:

* Male Age 45 or older
* Histologically confirmed adenocarcinoma of the prostate
* Disease Staging III or IV
* Clinical indication for androgen suppression therapy
* Serum testosterone at least 150 ng/dL at screening
* WHO Performance Scale 0 to 3
* Life expectancy of at least one year

Key Exclusion Criteria:

* Bilateral orchiectomy
* Prior androgen-ablative therapy within past year
* Second malignancy with 5 years (except adequately treated non-melanomatous skin cancer or superficial bladder cancer)
* Spinal cord compression

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2000-04; Primary Completion 2003-08 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Suppression of testosterone to chemical castration levels (<= 50 ng/dL) | 52 weeks

SECONDARY OUTCOMES:
PSA measurements | 52 weeks
Pain measurements | 52 weeks
QoL outcomes | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Regulatory Division, Study Director — Endo Pharmaceuticals (formerly Valera/Indevus Pharmaceuticals)

REFERENCES:
- [Result] Schlegel PN; Histrelin Study Group. Efficacy and safety of histrelin subdermal implant in patients with advanced prostate cancer. J Urol. 2006 Apr;175(4):1353-8. doi: 10.1016/S0022-5347(05)00649-X. PMID 16515997